CLINICAL TRIAL: NCT02676323
Title: A Phase I and Dose Expansion Cohort Study of Panobinostat in Combination With Fludarabine and Cytarabine in Pediatric Patients With Refractory or Relapsed Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: Panobinostat With Fludarabine and Cytarabine for Treatment of Children With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANAML; NCI-2016-00098 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Maximum tolerated dose; Childhood leukemia; Hematological malignancies
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Hematologic Neoplasms | interventions — Panobinostat; fludarabine; fludarabine phosphate; Cytarabine; Methotrexate; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants will be given panobinostat in combination with fludarabine and cytarabine. Treatment consists of one course of therapy given over 12 days. Participants will also receive intrathecal triples and leucovorin
  Interventions: Drug: Panobinostat; Drug: Fludarabine; Drug: Cytarabine; Drug: Intrathecal Triples; Drug: Leucovorin

INTERVENTIONS:
Drug: Panobinostat — Panobinostat will be given orally (PO) on days 1, 3, 5, 8, 10, and 12.
  Other Names: LBH589
Drug: Fludarabine — Fludarabine will be given intravenously (IV), 30 mg/m^2/dose over 30 minutes, daily for 5 days (days 8-12).
  Other Names: Fludara®; Fludarabine phosphate; 2-fluoro-ara-AMP
Drug: Cytarabine — Cytarabine will be given IV, 2 gram/m^2/dose over 4 hours, daily for 5 days (days 8-12).
  Other Names: Cytosine arabinoside; Ara-C; Cytosar®
Drug: Intrathecal Triples — Given intrathecally (IT).
  Other Names: ITMHA; methotrexate/hydrocortisone/cytarabine
Drug: Leucovorin — Leucovorin (5 mg/m^2/dose, max 5 mg) may be given PO or IV at 24 and 30 hours after each ITMHA.
  Other Names: Leucovorin calcium; Leucovorin rescue

SUMMARY:
Cancer is the uncontrolled growth of human cells. The growth of normal human cells is controlled by multiple mechanisms. Panobinostat belongs to a class of chemotherapy drugs called "histone deacetylase (HDAC) inhibitors." HDAC inhibitors like panobinostat block enzymes known as histone deacetylases, which stops cancer cells from dividing and causes them to die. Fludarabine and cytarabine are chemotherapy drugs that are commonly used to treat pediatric patients with refractory or relapsed acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS).

The purpose of this study is to test the safety of panobinostat and to find the highest dose of panobinostat that can be given safely when it is combined with fludarabine and cytarabine.

This pilot study will be done in two parts: The goal of Part 1 of the study is to find the highest tolerable dose of panobinostat that can be given to patients with AML or MDS, when it is combined with fludarabine and cytarabine. Once that dose is determined, participants will be enrolled on Part 2: Dose Expansion, to look at the effect of the panobinostat/fludarabine/cytarabine combination in patients with leukemia/MDS.

PRIMARY OBJECTIVE:

* Determine a tolerable dose of panobinostat when given in combination with fludarabine and cytarabine in pediatric patients with relapsed or refractory AML or MDS.

SECONDARY OBJECTIVES:

* Characterize the pharmacokinetics of panobinostat after the first dose and at steady-state.
* Estimate the overall response rate to the combination of panobinostat, fludarabine, and cytarabine.

DETAILED DESCRIPTION:
STUDY PART 1: Dose Escalation Cohort

During the dose escalation phase (Part 1), participants will receive one course of panobinostat plus fludarabine and cytarabine. The starting dose of panobinostat will be 10 mg/m^2/dose, with 2 additional dose levels of 15 and 20, depending on tolerability. Each course is 12 days

STUDY PART 2: Dose Expansion Cohort

The recommended phase 2 dose (RP2D) will be chosen based on the maximum tolerated dose (MTD) and the totality of data obtained from study Part 1. Additional patients will be enrolled, if needed, so that at least 6 patients are treated with the recommended RP2D to confirm the MTD of panobinostat to be given in study Part 2.

After final MTD determination, 12 additional participants will be treated at this dose level for further evaluation of tolerability and response, including more complete toxicity data and estimation of the response rate to the combination of panobinostat, fludarabine, and cytarabine.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of AML or MDS and must have disease that has relapsed or is refractory to chemotherapy, or that has relapsed after hematopoietic stem cell transplantation (HSCT).

  * Refractory disease is defined as persistent disease after at least two courses of induction chemotherapy.
  * Patients with AML must have ≥ 5% leukemic blasts in the bone marrow or increasing levels of minimal residual disease (MRD) in the bone marrow as assessed by flow cytometry. If an adequate bone marrow sample cannot be obtained, patients may be enrolled if there is unequivocal evidence of leukemia in the peripheral blood.
* Adequate organ function defined as the following:

  * Direct bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN
  * Creatinine ≤ 1.5 x ULN for age
  * Serum albumin > 3.0 g/dl
  * Left ventricular ejection fraction ≥ 40% or shortening fraction ≥ 25%.
* Age ≤ 24 years
* Patients must be able to swallow capsules
* Performance status: Lansky ≥ 50 for patients who are ≤ 16 years old and Karnofsky ≥ 50% for patients who are > 16 years old.
* Patients must have fully recovered from the acute effects of all prior therapy and must meet the following criteria:

  * At least 14 days must have elapsed since the completion of myelosuppressive therapy
  * At least 24 hours must have elapsed since the completion of low-dose chemotherapy, such as hydroxyurea or low-dose cytarabine (up to 200 mg/m^2/day).
  * For patients who have received prior HSCT, there can be no evidence of GVHD and greater than 60 days must have elapsed since the HSCT. Patients cannot be receiving therapy, including steroids, for the treatment or prevention of GVHD. All such medications must be discontinued at least 24 hours prior to enrollment.
* Body Surface Area: Because the smallest capsule size available for the panobinostat is 10 mg, the minimum BSA allowed for enrollment at Dose Level 1 to 0.85 m^2. The minimum for Dose Level 2 is BSA=0.6 m^2 and the minimum for Dose Level 3 is BSA=0.42 m^2.

Exclusion Criteria:

* Must not be pregnant or breastfeeding. Female patients who are sexually active and of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients who are sexually active must use an effective barrier method of contraception if sexually active with a female of child-bearing potential. For both male and female patients who are sexually active, effective methods of contraception must be used throughout the study and for three months following the last dose. Abstinence is an acceptable form of contraception.
* Patients with Down syndrome, acute promyelocytic leukemia, juvenile myelomonocytic leukemia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or other bone marrow failure syndromes are not eligible.
* Use of investigational agents within 30 days.
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, study participation, follow up, or interpretation of study research.
* Uncontrolled infection within one week of the first dose. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable.
* Known human immunodeficiency virus infection (pre-study testing not required).
* Patient with diarrhea > CTCAE grade 2. (CTCAE version 4.0)
* Impaired cardiac function or clinically significant cardiac diseases, history of arrhythmia (including ventricular fibrillation or torsade de pointes), bradycardia <50 bpm, screening ECG with prolonged QTc (> 450 msec), uncontrolled hypertension or any history or presence of sustained ventricular tachyarrhythmia.
* Impairment of GI function or GI disease that may significantly alter the absorption of panobinostat.
* Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting treatment. Granisetron may be administered, but antiemetics associated with QT prolongation (e.g., ondansetron) are not allowed.

Max Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 56 days following first dose of panobinostat
  Any participant who experiences non-hematologic dose-limiting toxicity (DLT) during the first 28 days after taking the initial dose of panobinostat and before receiving non-protocol therapy is considered evaluable for toxicity. Non-hematologic DLT includes any Grade 5 event and any Grade 3 or 4 event that is at least possibly related to panobinostat, unless the event is clearly due to extraneous causes or disease progression. Hematologic DLT includes failure to recover counts by Day 56 in the absence of persistent leukemia.
  Participants without DLTs who receive at least 5 of the 6 prescribed cycle I doses of panobinostat and can be followed for 28 days (56 days for evaluation of hematologic toxicity) after their initial dose of panobinostat are considered evaluable for toxicity. Participants who are not evaluable for toxicity will be replaced.
  The MTD is defined as the highest dose level at which six participants have been treated with at most one participant experiencing a DLT.

SECONDARY OUTCOMES:
Clearance (CL) | From baseline pre-dose day 1 through 48 hours after panobinostat administration
  Plasma samples will be analyzed via a validated method for plasma panobinostat concentration. Panobinostat concentration data will be analyzed in a non-linear mixed effects population pharmacokinetic (PK) model to determine the clearance.
Clearance (CL) | On day 8 from pre-dose through 48 hours after panobinostat administration
  Plasma samples will be analyzed via a validated method for plasma panobinostat concentration. Panobinostat concentration data will be analyzed in a non-linear mixed effects population pharmacokinetic (PK) model to determine the clearance.
Drug Absorption (ka) | From baseline pre-dose day 1 through 48 hours after panobinostat administration
  Plasma samples will be analyzed via a validated method for plasma panobinostat concentration. Panobinostat concentration data will be analyzed in a non-linear mixed effects population pharmacokinetic (PK) model to determine the drug absorption.
Drug Absorption (ka) | On day 8 from pre-dose through 48 hours after panobinostat administration
  Plasma samples will be analyzed via a validated method for plasma panobinostat concentration. Panobinostat concentration data will be analyzed in a non-linear mixed effects population pharmacokinetic (PK) model to determine the drug absorption.
Area under curve (AUC) | From baseline pre-dose day 1 through 48 hours after panobinostat administration
  Plasma samples will be analyzed via a validated method for plasma panobinostat concentration. Panobinostat concentration data will be analyzed in a non-linear mixed effects population pharmacokinetic (PK) model to determine the PK parameters. The AUC will be estimated based on the individual estimated PK.
Area under curve (AUC) | On day 8 from pre-dose through 24 hours after panobinostat administration
  Plasma samples will be analyzed via a validated method for plasma panobinostat concentration. Panobinostat concentration data will be analyzed in a non-linear mixed effects population pharmacokinetic (PK) model to determine the PK parameters. The AUC will be estimated based on the individual estimated PK.
Maximum concentration (Cmax) | From baseline pre-dose day 1 through 48 hours after panobinostat administration
  Plasma samples will be analyzed via a validated method for plasma panobinostat concentration. Panobinostat concentration data will be analyzed in a non-linear mixed effects population pharmacokinetic (PK) model to determine the PK parameters. The Cmax will be estimated based on the individual estimated PK.
Maximum concentration (Cmax) | On day 8 from pre-dose through 24 hours after panobinostat administration
  Plasma samples will be analyzed via a validated method for plasma panobinostat concentration. Panobinostat concentration data will be analyzed in a non-linear mixed effects population pharmacokinetic (PK) model to determine the PK parameters. The Cmax will be estimated based on the individual estimated PK.
Complete response (CR) rate | Up to Day 42 after completion of therapy
  Response will be based on blast percentage by flow cytometry. Blast percentages determined by morphology will be used in cases that are not evaluable by flow cytometry.
  The efficacy of the combination of panobinostat and chemotherapy, as measured by the CR rate will be assessed for patients enrolled at the MTD. The rate of CR will be presented as a point estimate with a 95% exact binomial confidence interval.
Overall response (OR) rate | Up to Day 42 after completion of therapy
  Response will be based on blast percentage by flow cytometry. Blast percentages determined by morphology will be used in cases that are not evaluable by flow cytometry.
  The efficacy of the combination of panobinostat and chemotherapy, as measured by the OR (CR + incomplete blood count recovery + partial response + therapeutic success) will be assessed for the patients enrolled at the MTD. The rate of OR will be presented as a point estimate with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E. Rubnitz, MD,PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (7):
- United States (7):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital and Health Center, San Diego, California
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols